CLINICAL TRIAL: NCT01802060
Title: Accuracy of SPD Persona LH Assay When Compared to Ultrasound Observed Ovulation and Other Indices of Ovulation
Status: Completed | Type: Observational
Sponsor: SPD Development Company Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: PROTOCOL-0449
Record Dates: First submitted 2013-01-29; First posted 2013-03-01 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Ovulation
Keywords: Persona; E3G; LH; ovulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine samples Serum samples
Oversight: Data Monitoring Committee: No

SUMMARY:
This study will examine the performance of the Persona assays in identifying the time when risk of pregnancy is highest by comparing results to ultrasound observed ovulation and other indices of ovulation.

DETAILED DESCRIPTION:
Persona is a CE marked, natural method of contraception that works by monitoring hormone changes in a woman's urine to identify the days of her menstrual cycle when she is likely to become pregnant following unprotected intercourse. Persona consists of test sticks that measure luteinising hormone (LH) and estrone-3-glucuronide (E3G), which are read by a handheld monitor. This hormonal data is converted using a proprietary algorithm, into simple-to-understand information on the user's contraceptive status; a "red light" where she needs to abstain from intercourse to avoid pregnancy, or a "green light" where unprotected intercourse is unlikely to lead to pregnancy. A prospective 13 cycle reliability study has found Persona to be 94% effective.

This study will examine the relationship between the information provided by the Persona assays and ultrasound observed ovulation, along with other indicators of when a woman is fertile (basal body temperature (BBT) measurement and cervical secretion observations).

This is a single centre clinical study which will be conducted at the green-ivf clinic in Grevenbroich, Germany. The primary objective will be to assess the difference between the timing of the LH surge detected by Persona and observed ovulation by reference to transvaginal ultrasound examination.

In addition, comparison of Persona determined levels of LH and E3G will be made to urine and serum levels of these and other reproductive hormones. Comparison will also be made to BBT and cervical secretion observations which are indirect measurements of the fertile phase.

In order to achieve these objectives, a minimum of 40 female volunteers will be recruited by the study site either out of the patient pool coming for routine gynaecological examination or from the general population via newspaper advertisement.

The study will last for one menstrual cycle starting on the first day of menstrual bleeding (day 1 of the cycle) and concluding with the onset of the next menses. Volunteers will be asked to collect daily urine samples and use an adapted Persona monitor for the duration of the study as per the first cycle of use (i.e. a maximum of 16 tests). The monitor will be adapted to blind the user from the result of each test. Volunteers will therefore be advised that the modified Persona monitor cannot be used as a contraceptive device during the study. Volunteers will also be asked to take daily measurements of BBT and to record this along with cervical secretion observations on a daily natural family planning (NFP) chart.

Volunteers will be required to attend for a recruitment visit to the trial site followed by approximately 12 visits either daily, or two days apart. Transvaginal ultrasonography will be carried out on cycle days 5, 7, 9, 11 and daily from 16mm follicular size onwards until ovulation has occurred. Blood sampling will also be conducted on these days as well as on day 7 and day 9 post-ovulation.

Ultrasound examinations, blood sampling and hormonal blood tests will be performed at the trial centre. Urine samples will be shipped to the study sponsor for hormonal analysis.

Diary and scan data will also be transferred to the study sponsor to provide a single data set for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Aged 18 - 40 years
* Menstrual cycle length between 23 and 35 days
* Had two natural cycles prior to study participation
* Using non-hormonal contraception to avoid pregnancy OR abstaining from intercourse for the last three months and the present cycle

N.B: Non hormonal contraception includes barrier methods such as male and female condoms, diaphragms or caps, non-hormonal intra-uterine devices such as coils, male and female sterilisation or natural family planning

Exclusion Criteria:

* Unwilling to provide written informed consent to participate in the study or comply with study procedures
* Pregnant
* Breastfeeding
* Has menopausal symptoms such as night sweats or hot flushes
* Using any hormonal treatments e.g. hormonal contraception, fertility treatments and hormone replacement therapy (except thyroxin)
* Taking antibiotics (based on decision by principle investigator)
* Has a diagnosis of polycystic ovarian syndrome (PCOS)
* Has impaired liver or kidney function
* Intending to use PERSONA as a contraceptive during the study period
* Contraindications to frequent blood sampling e.g. anaemia, hypotonia and blood clotting diseases
* Contraindications to frequent ultrasound examinations e.g. morbid obesity and recent abdominal surgery

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: General Public
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2013-02; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Ultrasound | Participants will be followed for one menstrual cycle, anticipated average of four weeks.
  Accuracy of the LH urine assay contained within PERSONA at predicting ovulation, by comparing the day of the LH surge with ultrasound observed ovulation

SECONDARY OUTCOMES:
Quantitative determination of urinary and serum levels of LH and E3G | Participants will be followed one menstrual cycle, an anticipated four weeks
  Comparison of Persona determined levels of LH and E3G will be made to urine and serum levels of these and other reproductive hormones.
Volunteer recorded BBT and cervical secretion observations. | Participants will be followed for one menstrual cycle, an anticipated four weeks
  Comparison of Persona determined levels of LH and E3G will be made to BBT and cervical secretion observations which are indirect measurements of the fertile phase.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Gnoth, Dr, Principal Investigator — Green-ivf, Rheydter Strasse 143
Locations (1):
- Green-ivf, Rheydter Strasse 143, Grevenboich, Düsseldorf, Germany

REFERENCES:
- [Derived] Gnoth C, Roos J, Broomhead D, Schiffner J, Godehardt E, Freundl G, Johnson S. Antimullerian hormone levels and numbers and sizes of antral follicles in regularly menstruating women of reproductive age referenced to true ovulation day. Fertil Steril. 2015 Dec;104(6):1535-43.e1-4. doi: 10.1016/j.fertnstert.2015.08.027. Epub 2015 Sep 15. PMID 26384163
- [Derived] Johnson S, Weddell S, Godbert S, Freundl G, Roos J, Gnoth C. Development of the first urinary reproductive hormone ranges referenced to independently determined ovulation day. Clin Chem Lab Med. 2015 Jun;53(7):1099-108. doi: 10.1515/cclm-2014-1087. PMID 25720077